CLINICAL TRIAL: NCT02464475
Title: Effects of Osteopathic Manual Treatment on Interoception: 2- Armed RCT on cLBP Patients
Brief Title: Effects of OMT on Interoception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Come Collaboration (Other)
Collaborators: University of Chieti (Other)
Responsible Party: Principal Investigator, Francesco Cerritelli, DO, MS, Come Collaboration
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: InterOST
Record Dates: First submitted 2015-05-28; First posted 2015-06-08 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Chronic Low Back Pain
Keywords: osteopathic manipulative treatment; interoception
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OMT (Experimental)
  Interventions: Other: osteopathic manipulative treatment
- Sham (Sham Comparator)
  Interventions: Other: sham osteopathic treatment

INTERVENTIONS:
Other: osteopathic manipulative treatment
  Arms: OMT
Other: sham osteopathic treatment
  Arms: Sham

SUMMARY:
Recent evidence suggested that the anterior insula cortex seems to be the main site of interoception. Several studies showed an association between change in insula function and interoception, bodily perception and consciousness in subjects with chronic pain. Although osteopathic research has been demonstrated to be effective in reducing pain, studies exploring the effect of osteopathy on interoception are lacking. Therefore, the aim of the present study is to explore the extent to which osteopathic treatment could modify interoception parameters both measuring brain functional connectivity and clinical questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain
* written informed consent signed

Exclusion Criteria:

* congenital disease
* acute pain
* subject below 30 and above 50
* co-morbidities associated with low back pain
* surgical patients
* cardio-vascular, respiratory, gastro-enteric disease
* obese subjects
* diabetics
* dizziness
* subjects into pharmacological prophylaxis
* drug addicted subjects
* subjects undergoing physiotherapy
* subjects with experience in osteopathic treatment

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
functional connectivity on right anterior insula cortex | 4 weeks
  before-after change in fMRI values

SECONDARY OUTCOMES:
differences on salience network activities | 4 weeks
  report any change between study and control group on pattern activation of salience network
acute changes on salience network | 2 hours
  voxel differences
resting state network differences between groups | 4 weeks
  voxel differences
DTI changes between groups | 4 weeks
  differences in DTI parameters and indexes
changes in GABA concentration | 4 weeks
  amount of GABA in the given voxel
changes in quality of life | 4 weeks
  SF-36v2 self-reported questionnaire
changes in perception of pain | 4 weeks
  McGill self-reported questionnaire
changes in disability | 4 weeks
  Oswestry disability questionnaire
changes in depression symptoms | 4 weeks
  Beck Depression Inventory questionnaire
changes in anxiety symptoms | 4 weeks
  Hospital Anxiety and Depression Scale questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Cerritelli, MS, DO, Principal Investigator — University of Chieti-Pescara
Locations (1):
- University of Chieti-Pescara, Chieti, Italy